CLINICAL TRIAL: NCT06496412
Title: Safety and Efficacy of Fecal Microbiota Transplantation on Cognitive Function in T1DM: a Randomized Controlled, Triple-blind Clinical Study
Brief Title: Safety and Efficacy of Fecal Microbiota Transplantation on Cognitive Function in T1DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Xia Li, Professor, Department of Endocrinology, Institute of of Metabolism and Endocrinology, National Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital of Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T1D cognitive impairment FMT
Record Dates: First submitted 2024-06-25; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; fecal microbiota transplantation; cognitive impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cognitive Dysfunction | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fecal microbiota transplantation (Experimental): On the basis of baseline medication, high-dose fecal microbiota transplantation (FMT) will be administered, with subjects taking 50 fecal microbiota capsules. Subsequently, maintenance doses will be administered at week 2, 4, 8, 12, and 20, with 10 capsules taken each time. Fasting is required 4 hours before and 1 hour after capsule ingestion, and subjects are instructed to maintain a stable diet and physical activity pattern throughout the 24-week study period. Capsules will be transported on ice and warmed for 10 minutes at 37°C before FMT administration.
  Interventions: Drug: fecal microbiota transplantation
- placebo (Placebo Comparator): Different from the experimental group, the control group will receive placebo capsules that have the same appearance as the fecal microbiota capsules, while other procedures remain the same as those in the experimental group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fecal microbiota transplantation — Take fecal microbiota capsules.
  Arms: fecal microbiota transplantation
Drug: Placebo — Take placebo capsules.
  Arms: placebo

SUMMARY:
This study is a prospective, single-center, parallel-design,1:1 randomized controlled trial with triple blinding. It aims to investigate the effects of fecal microbiota transplantation (FMT) on cognitive function in patients with long-term type 1 diabetes (T1D), as well as its effects on other complications, glycemic control, insulin dosage, insulin resistance, peripheral blood immune cells, serum metabolites, and safety. This study is divided into two phases for recruiting participants. The first phase recruits 10 individuals (experimental group: 5, control group: 5), while the second phase recruits 30 individuals (experimental group: 15, control group: 15).The main research objectives are as follows:

1. To observe the difference in cognitive function between the FMT group and the placebo group, with the indicators including cognitive scale scores, changes in brain MRI imaging indicators and brain age at week 24 compared to baseline.
2. To observe the difference in other complications between the FMT group and the placebo group, with the indicators including changes in urinary albumin/creatinine ratio, fundus photography, carotid intima-media thickness, and arterial pulse wave velocity at week 24 compared to baseline.
3. To observe the difference in glycemic control, insulin dosage, insulin resistance, peripheral blood immune cells, gut microbiota, and serum metabolites between the FMT group and the placebo group.
4. To evaluate the safety of FMT.

ELIGIBILITY:
Inclusion Criteria:

1. According to the definition of type 1 diabetes mellitus (T1DM) by the World Health Organization (WHO), the diagnostic criteria are as follows: (i) clinically diagnosed as T1D by endocrinologists; (ii) insulin dependence from disease onset and diabetic ketoacidosis (DKA)/diabetic ketosis (DK) at diagnosis; (iii) positive for at least one of islet autoantibodies for glutamic acid decarboxylase antibody [GADA], insulinoma-associated protein 2 antibody [IA-2A], and zinc transporter 8 antibody [ZnT8A]; or negative for all three islet autoantibodies, but diagnosed before age 30.
2. Age between 18 and 60 years, with a diabetes duration of 10 years or more
3. Glycated hemoglobin levels ranging from 6.5% to 9.0%.

Exclusion Criteria:

1. Use of any hypoglycemic medication other than insulin in the two months prior to randomization.
2. Participation in other clinical trials within the two months prior to randomization.
3. Use of antimicrobial drugs, probiotics, intestinal microbiota regulators, and other drugs with significant impact on gut microbiota within the two months prior to randomization.
4. Gastrointestinal diseases: celiac disease, irritable bowel syndrome, Crohn's disease, etc.
5. Severe infections, severe heart, liver, kidney diseases, tumors, and other inflammatory or autoimmune diseases.
6. Pregnant or lactating women, or women planning pregnancy during the study period.
7. Severe mental health disorders such as schizophrenia, major depression, bipolar disorder, alcohol or substance abuse, etc.
8. Neurological disorders such as Parkinson's disease, progressive supranuclear palsy, epilepsy, multiple sclerosis, traumatic brain injury, stroke, etc.
9. Post-implantation of metal materials or contraindications for other MRI examinations.
10. Severe episodes of unconscious hypoglycemia within the past two months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Cognition:Comparison of the average change in Z-scores for memory and executive domain-related assessments between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Z-scores of memory and executive domain assessments-related assessments are indicators that can comprehensively reflect cognitive function.
Cognition: Comparison of the average change in Auditory Verbal Learning Test between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Auditory Verbal Learning Test (AVLT) is a neuropsychological assessment tool used to evaluate an individual's verbal learning and memory skills. This test involves the presentation of a list of words to the test subject, who is then asked to recall as many words as possible from the list after a single exposure. The process is typically repeated several times, allowing the examiner to assess the subject's ability to learn new information and retain it over time.
Cognition: Comparison of the average change in Trail Making Test Part A and Part B between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts, A and B. Participant is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Cognition: Comparison of the average change in Verbal Fluency Test between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Verbal Fluency Test (VFT) is a common neuropsychological assessment used to evaluate an individual's cognitive flexibility and generative language abilities. It typically involves asking the participant to produce as many words as possible within a certain time limit, usually one minute, that fit a specific criterion.
Cognition: Comparison of the average change in Boston Naming Test between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Boston Naming Test (BNT) is a widely used neuropsychological instrument designed to assess an individual's confrontational naming abilities, which is a critical aspect of language function. The test consists of a series of line drawings of objects, animals, and people, each paired with a prompt that encourages the participant to name the item.
Cognition: Comparison of the average change in Stroop Color- Word Association Test between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Stroop Color- Word Association Test is particularly useful in assessing executive functions, such as selective attention and cognitive flexibility. It is sensitive to the effects of various conditions that impact cognitive control, including attention deficit hyperactivity disorder (ADHD), Alzheimer's disease, Parkinson's disease, and substance abuse disorders. The test can also be used to evaluate the effectiveness of cognitive training programs and to monitor changes in cognitive function over time.
Cognition: Comparison of the average change in Symbol Digit Modalities Test between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Symbol Digit Modalities Test (SDMT) is a brief neuropsychological screening tool designed to assess cognitive processing speed and attention. The SDMT is scored based on the number of correct responses within the time frame, providing a quantitative measure of cognitive performance. It is particularly sensitive to changes in cognitive function that may occur with aging, as well as in conditions such as multiple sclerosis, Parkinson's disease, traumatic brain injury, and Alzheimer's disease. The test is often used to monitor the progression of cognitive decline and to evaluate the effectiveness of treatments.
  The SDMT is also valuable in differentiating between different types of cognitive impairments and can be used as part of a comprehensive neuropsychological assessment to provide a more detailed picture of an individual's cognitive strengths and weaknesses. Its brevity and ease of administration make it a practical tool for repeated assessments over time.
Cognition: Comparison of the average change in Clock drawing test between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Clock Drawing Test (CDT) is a widely used neuropsychological screening tool that assesses an individual's cognitive function, particularly in the areas of executive function, visual-spatial skills, and constructional praxis. It is a simple yet effective test that requires participants to draw a clock face and then set the hands to indicate a specific time, often 10 minutes past 11.
Cognition: Comparison of the average change in MOCA between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Montreal Cognitive Assessment (MOCA) is a rapid screening tool for mild cognitive dysfunction, particularly useful in identifying early signs of cognitive impairment associated with conditions such as Alzheimer's disease and other forms of dementia.The test is sensitive to changes in cognitive function that may not be detected by less detailed assessments, making it a valuable tool for both clinical and research settings.
Cognition: Comparison of the average change in Subjective Cognitive Decline 9 between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Subjective Cognitive Decline 9 (SCD9) is a tool designed to assess an individual's perception of changes in their cognitive abilities over time. It is particularly useful for identifying early signs of cognitive decline that may be indicative of the onset of neurodegenerative diseases such as Alzheimer's disease.
  The development of the SCD9 questionnaire aims to provide a localized, sample-assisted, multi-domain instrument that can be used to evaluate subjective cognitive decline in the elderly population over the past 1-2 years. The scale has demonstrated good reliability and validity, with a confirmatory factor analysis supporting a 4-factor model that includes memory, attention, executive function, and language domains.
Cognition: Comparison of the average change in Brain MRI between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Brain MRI, particularly structural Structural MRI, Diffusion MRI(DTI), and Functional MRI (fMRI), plays a crucial role in understanding cognitive functions. Structural MRI can identify anatomical correlates of cognitive deficits, while DTI provides insights into the integrity of neural pathways essential for cognitive processing. fMRI allows researchers to observe brain activity during various cognitive tasks, offering a direct link between brain function and cognition. This comprehensive approach enables clinicians and researchers to explore the neural basis of cognitive functions and disorders, enhancing diagnosis and treatment strategies.

SECONDARY OUTCOMES:
Safety: Proportion of participants with treatment-related adverse events, serious adverse events, or adverse events of special interest. | from baseline to week 24
  Proportion of participants with treatment-related adverse events, serious adverse events, or adverse events of special interest.
  Adverse events, serious adverse events, or adverse events of special interest, will be evaluated following study procedures using AE and SAE forms, telephone and in person interview, and relevant medical records related to adverse events.
macrovascular complications：Comparison of the average change in Carotid Intima-Media Thickness between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Carotid Intima-Media Thickness is a valuable indicator of subclinical atherosclerosis and a predictor of cardiovascular and cerebrovascular events. It is typically measured using high-resolution B-mode ultrasonography, which provides images of the carotid artery walls. The measurement is taken from the leading edge of the lumen-intima interface to the leading edge of the media-adventitia interface on the far wall of the carotid artery.
macrovascular complications：Comparison of the average change in Arterial Pulse Wave Velocity between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Arterial Pulse Wave Velocity (PWV) is a measure of the speed at which blood pressure waves move through the arteries. It is an important indicator of arterial stiffness, with higher values indicating stiffer arteries, which are often associated with cardiovascular risk.
macrovascular complications：Comparison of the average change in Ankle-Brachial Index between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Ankle-Brachial Index (ABI) is a simple, non-invasive test used to assess the presence of peripheral artery disease (PAD). It compares the blood pressure measured at the ankle with the blood pressure measured at the arm (brachial artery).
  ABI is also a marker for overall cardiovascular health. A low ABI is associated with an increased risk of heart attack, stroke, and overall cardiovascular mortality.
microvascular complications：Comparison of the average change in Albumin-to-Creatinine Ratio between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Albumin-to-Creatinine Ratio (ACR) is a diagnostic test used to detect and monitor kidney function, particularly to identify early signs of kidney damage. It measures the amount of albumin (a type of protein) in the urine, normalized to the amount of creatinine (a waste product of muscle metabolism) to account for variations in urine concentration.
microvascular complications：Comparison of the average change in Estimated Glomerular Filtration Rate between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Estimated Glomerular Filtration Rate (eGFR) is a key indicator of kidney function. It estimates the rate at which the kidneys filter waste products from the blood, providing valuable information about renal health and helping to diagnose and monitor kidney disease.
microvascular complications：Compare the differences in the proportion of abnormal fundus photography and the severity of progression between the experimental and control groups during the follow-up period. | from baseline to week 24
  Fundus photography is a non-invasive diagnostic procedure used to capture images of the retina at the back of the eye. This technique is essential for the early detection, evaluation, and monitoring of diabetic retinopathy and other vascular changes in the eye, which can be indicative of diabetes-related complications.
microvascular complications：Comparison of the average change in Neuropathy lmpairment Score in the Lower Limbs between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Neuropathy Impairment Score in the Lower Limbs (NIS-LL) is a clinical tool used to evaluate the severity of neuropathy, specifically in the lower extremities. This score helps in assessing the degree of nerve damage and its impact on motor and sensory functions. The NIS-LL takes into account the following components.
Glycemic control：Comparison of the average change in Hemoglobin A1c between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Hemoglobin A1c (HbA1c) is a blood test that measures the average level of blood glucose (sugar) over the past two to three months. It is a key indicator used to diagnose and manage diabetes.
Glycemic control：Comparison of the average change in Time in Range between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Time in Range (TIR) is a key metric used in Continuous Glucose Monitoring (CGM) to assess glycemic control in individuals with diabetes. It represents the percentage of time that a person's blood glucose levels stay within a target range over a specified period, typically 24 hours.
Glycemic control：Comparison of the average change in Time Above Range between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Time Above Range (TAR) is a crucial metric in Continuous Glucose Monitoring (CGM) used to evaluate how often an individual's blood glucose levels exceed a predefined upper limit. This metric helps in understanding hyperglycemia and its potential impact on health.
Glycemic control：Comparison of the average change in Time Below Range between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Time Below Range (TBR) is a critical metric in Continuous Glucose Monitoring (CGM) used to evaluate the duration that an individual's blood glucose levels fall below a predefined lower limit. This metric is crucial for understanding hypoglycemia and its potential risks.
Glycemic control：Comparison of the average change in Glucose Management Indicato between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Glucose Management Indicator (GMI) is a metric used in Continuous Glucose Monitoring (CGM) to estimate average blood glucose levels over a specified period. It provides a simplified interpretation of glycemic control based on CGM data.
Glycemic control：Comparison of the average change in Glycemia risk index between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Glycemia risk index (GRI), a newly developed composite CGM metric, could evaluate the quality of glycemia by weighting the risk of both hypoglycemia and hyperglycemia, which are associated with long-term complications
Glycemic control：Comparison of the average change in Coefficient of Variation between the experimental and control groups from baseline to week 24. | from baseline to week 24
  The Coefficient of Variation (CV) in Continuous Glucose Monitoring (CGM) is a statistical measure used to assess the variability of blood glucose levels over a period of time. It provides insights into the stability and consistency of glucose control.
Glycemic control：Comparison of the average change in Mean Amplitude of Glycemic Excursions between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Mean Amplitude of Glycemic Excursions (MAGE) is a metric used in Continuous Glucose Monitoring (CGM) to quantify the magnitude of glucose fluctuations over a specified period. It provides insights into the variability and stability of blood glucose levels, reflecting how much and how often glucose levels deviate from a baseline.
Blood lipid：Comparison of the average change in triglycerides between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Triglycerides (TG) are the most common form of fat in the human body and serve as an important source of energy. They are a type of lipid, which is a waxy-like fat substance made by the body and obtained from foods that contain fat.
Blood lipid：Comparison of the average change in total cholesterol between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Total Cholesterol (TC) ,which stands for Total Cholesterol, is a blood test that measures the total amount of cholesterol in your blood. Cholesterol is a waxy substance that's vital for the body to function properly. However, too much cholesterol in your blood can lead to health problems, such as heart disease and stroke.
Blood lipid：Comparison of the average change in high-density lipoprotein cholesterol between the experimental and control groups from baseline to week 24. | from baseline to week 24
  High-Density Lipoprotein Cholesterol（HDL-C)）is commonly referred to as "good" cholesterol because high levels of HDL-C are associated with a lower risk of heart disease. HDL-C helps transport cholesterol from other parts of your body back to your liver, where it can be removed from your bloodstream. This process helps keep cholesterol from building up in your arteries, thus reducing the risk of atherosclerosis (hardening or narrowing of the arteries) and cardiovascular events such as heart attacks and strokes. Regular physical activity, a healthy diet, and certain medications can help increase HDL-C levels.
Blood lipid：Comparison of the average change in low-density lipoprotein cholesterol between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Low-Density Lipoprotein Cholesterol (LDL-C) is often referred to as "bad" cholesterol because high levels of LDL-C can lead to the buildup of cholesterol in the arteries, which increases the risk of atherosclerosis (hardening or narrowing of the arteries) and cardiovascular diseases such as heart attacks and strokes. LDL-C transports cholesterol from the liver to various parts of the body. If there is too much LDL-C in the blood, it can deposit on the walls of the arteries, forming plaques that can restrict or block blood flow. Managing LDL-C levels through diet, exercise, and medications is important for cardiovascular health.
Blood pressure：Comparison of the average change in blood pressure between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Blood pressure is the force exerted by circulating blood on the walls of the arteries. It is an essential measure of cardiovascular health and is typically recorded as two numbers: systolic and diastolic pressure.
  Systolic Pressure: The higher number, representing the pressure in the arteries when the heart beats and pumps blood.
  Diastolic Pressure: The lower number, representing the pressure in the arteries when the heart is at rest between beats.
Body Mass Index：Comparison of the average change in body mass index between the experimental and control groups from baseline to week 24. | from baseline to week 24
  Body Mass Index (BMI) is a widely used measure to assess whether a person has a healthy body weight for a given height. It is a simple calculation that provides an indication of body fatness, which can be related to the risk of developing health problems.
Insulin resistance: Comparison of the average change in estimated Glucose Disposal Rate between the experimental and control groups from baseline to week 24. | from baseline to week 24
  eGDR stands for "estimated Glucose Disposal Rate." It is a metric used to estimate insulin sensitivity, particularly in individuals with diabetes, especially type 1 diabetes. Insulin sensitivity refers to how effectively the body's cells respond to insulin, which is crucial for regulating blood glucose levels.
Insulin dose: Comparison of the average change in insulin dose between the experimental and control groups from baseline to week 24. | from baseline to week 24
  An insulin dose refers to the specific amount of insulin administered to a person with diabetes to help manage their blood glucose levels.
Change in gut composition: Engraftment of fecal microbial transplant as assessed by 16S rRNA sequencing of recipient stool sample | from baseline to week 24
  In order to determine efficacy of fecal transplant, change in composition, i.e. microbial engraftment will be assessed by testing for newly detected operational taxonomic units (OTUs) in the gut microbiome of a participant post-FMT (which were present in the donor but undetected in the participant pre-FMT). This will be assessed via 16S rRNA seq of recipient stool samples pre- and post- FMT.
Changes in peripheral blood mononuclear cells: Assessing the effects of fecal microbial transplant on peripheral blood mononuclear cells by flow cytometry. | from baseline to week 24
  Flow cytometry is a powerful technique used to analyze the characteristics of individual cells in a heterogeneous population. When applied to peripheral blood mononuclear cells (PBMCs), flow cytometry provides detailed insights into the composition and function of various immune cell subsets present in the bloodstream.
Changes in peripheral blood metabolites: Assessing the impact of fecal microbiota transplantation on peripheral blood metabolites using metabolomics. | from baseline to week 24
  Metabolomics is a powerful analytical approach used to comprehensively analyze and quantify small molecules, known as metabolites, present in biological samples. When applied to peripheral blood, metabolomics enables the identification and measurement of a wide range of metabolites that serve as indicators of various physiological processes and metabolic pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Li, MD/PHD, Principal Investigator — The Second Xiangya Hospital, Central South University
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No